CLINICAL TRIAL: NCT06077539
Title: Dexmedetomidine Versus Ketamine Versus Magnesium Sulfate for the Prevention of Emergence Agitation Following Sevoflurane Induced Anesthesia in Cardiac Catheterization in Pediatrics : A Prospective, Double-blinded, Randomized Controlled Study.
Brief Title: Dexmedetomidine Versus Ketamine Versus Magnesium Sulfate for the Prevention of Emergence Agitation Following Sevoflurane Induced Anesthesia in Cardiac Catheterization in Pediatrics
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Assistant professor of anesthesia ,surgical intensive care and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: N-122-2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Ketamine; Magnesium; Saline Solution

STUDY DESIGN:
Intervention Model Description: (100) patients will be randomized into four equal groups using computer-generated block randomization and there will be five blocks each block contains 5 patients in each group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist not involved in the study will open envelopes and will prepare the drug. All syringes will be prepared by the same investigator not one of the study researchers. Administration of anesthesia and study drugs will be made by other investigators blinded to the study drugs and not involved in the study. Data collection will be done by investigator who is included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine group (Active Comparator): 25 patients will receive Dexmedetomidine 1 μg/kg bolus over 10 min followed by 0.5 μg/kg/h as maintenance volume-matched 0.9% saline.
  Interventions: Drug: Dexmedetomidine
- Magnesium group (Active Comparator): 25 patients will receive IV magnesium as a loading dose 15 mg/kg diluted in 0.9% NaCl given over 10 min followed by 10mg/kg/h IV infusion( for Concentration of solution will not exceed 1gm/25 mL (40 mg/ml).
  Interventions: Drug: Magnesium
- Ketamine group (Active Comparator): 25 patients will receive intravenous (IV) ketamine 1mg/kg diluted in 0.9% NaCl as a loading dose over 10min then 1mg/kg/h IV infusion
  Interventions: Drug: Ketamine
- Control group (Placebo Comparator): in 25 patients saline will be given as bolus over 10 min then will be infused as maintenance by the same rate of the other groups.
  Interventions: Other: normal saline 0.9% NaCL

INTERVENTIONS:
Drug: Dexmedetomidine — a selective a-2 adrenoceptor agonist, has sedative, analgesic, and anxiolytic effects.
  Arms: Dexmedetomidine group
Drug: Ketamine — NMDA (N-methyl-D-aspartate) receptor antagonist
  Arms: Ketamine group
Drug: Magnesium — NMDA (N-methyl-D-aspartate) receptor antagonist
  Arms: Magnesium group
Other: normal saline 0.9% NaCL — saline will be given as bolus over 10 min then will be infused as maintenance by the same rate of the other groups
  Arms: Control group

SUMMARY:
Emergence agitation (EA) is a post-operative behavioral disturbance was first reported in early 1960s. EA is a term used to describe non purposeful restlessness and agitation, thrashing, crying or moaning, disorientation and incoherence during early stage of recovering from general anesthesia in children, especially those receiving sevoflurane. Generally, the incidence of EA following sevoflurane anesthesia varies from 10% to 66% and is more common in pre-school children. EA is generally short lived without obvious aftereffect. However, it still accompanies with risk of self-injury, and requires extra nursing care, which may delay the discharge and increase the cost of medical care Emergence agitation is diagnosed by a final composite score of greater than or equal to 10 on the Pediatric Anesthesia Emergence Delirium Scale (PAED).(

DETAILED DESCRIPTION:
Sevoflurane induced anesthesia does not cause significant cardiac depression and dysrrhythmias as compared to halothane. Sevoflurane anesthesia is also easy to titrate for maintaining an adequate level of anesthesia, especially for the intubated. It also is a potent bronchodilator, which can offer an added benefit especially in children with a history of asthma. For all above reasons sevoflurane has clearly become the inhalation induction agent of choice.

The exact reasons for a higher incidence of EA with sevoflurane are not well explained. seizure activity in previously nonepileptic patients has been detected with electroencephalography during sevoflurane anesthesia.

One of the proposed treatments for EA is the use of opioids; however, it carries the risk of an extended Post Anesthetic Care Unit (PACU) stay resulting in parents' discomfort and added costs. Therefore, analgesic adjuvants with NMDA (N-methyl-D-aspartate) receptor antagonist functions, such as ketamine and magnesium sulfate have been tried to control this phenomenon in children.

Also, Dexmedetomidine, a selective a-2 adrenoceptor agonist, has sedative, analgesic, and anxiolytic effects. It was proved that α2 agonists decrease emergence agitation by their analgesic effect as well as by minimizing the anesthetic requirements.

In the review of literature this is the first study comparing the effectiveness of the three drugs ketamine, magnesium sulfate and dexmedetomidine infusions together in one study on the incidence of emergence agitation after sevoflurane induced anesthesia in children.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II
* ages from 2-5 years.
* weight more than 6 kg.
* scheduled for cardiac catheterization procedure not exceeding 3 hours.

Exclusion Criteria:

* psychological disorder or cognitive delay.
* chronic or acute intake of any sedative drug or anticonvulsant drugs.
* Any neurological condition that will limit ability to communicate with, or understand a practitioner.
* those with coexisting renal diseases , any reported allergy to the given medications.
* legal guardian refusal .

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
PAED scale 15 min postoperatively | 15 minutes
  pediatric anesthesia emergence delirium

CONTACTS AND LOCATIONS:
Overall Officials: Amany Saleh, MD, Principal Investigator — Cairo University
Locations (1):
- Amany Hassan Saleh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol